CLINICAL TRIAL: NCT02335034
Title: Project Osteoarthritis: Recovering Quality of Life by Means Education II (PARQVE II) - A Prospective Randomized Study Comparing the Multidisciplinary Care Associated With Education to Multidisciplinary Treatment Without Education.
Brief Title: Project Arthritis Recovering Quality of Life by Means Education II (PARQVE II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: TRB Chemedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12671/14
Record Dates: First submitted 2014-12-22; First posted 2015-01-09 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2019-01

CONDITIONS: Knee Osteoarthritis; Osteoarthritis
Keywords: Osteoarthritis; Knee; Education; Quality of life; Treatment outcome; Musculoskeletal pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Musculoskeletal Pain | interventions — Referral and Consultation

STUDY DESIGN:
Masking Description: single-blind
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): Intervention: study group will attend two days of classes (two months apart) with the seven professional teams, covering what is the disease arthritis, its causes and treatment options; what is disease, being ill, and the role of the patient in the treatment to obtain behavioral change; the importance of exercise in relieving symptoms, the importance of rest and proper ergonomics at home and at work; proper alimentation; the difference between labor work and regular physical activity as well as the importance of strength resistance and stretching exercises; and the importance of leisure. The second intervention verifies the acquired concepts.
  Interventions: Behavioral: Study Group Educational courses, DVD, print material of lectures
- Control Group (Experimental): The control group will only make evaluations / consultations with all professional teams without classes for 2 years, then will attend the courses and will be followed by two more years.
  Interventions: Behavioral: Control Group only make evaluations / consultations with all professional teams

INTERVENTIONS:
Behavioral: Study Group Educational courses, DVD, print material of lectures — 2 Educational courses (two months apart). Receive DVD and printed material of the lectures.
  Arms: Study group
Behavioral: Control Group only make evaluations / consultations with all professional teams — Evaluations and consultations with all professional teams without classes for 2 years.
  At two years: two days of lectures two months apart with DVD and printed material of the lectures. Will be followed by two more years.
  Arms: Control Group

SUMMARY:
OBJECTIVE: To evaluate the improvement of patients with gonarthritis exposed to a multidisciplinary care program with and without associated classroom educational program. METHODS: 152 patients (men and women) aged 40 or older with arthritis stages I to III of Kelgren and Lawrence. Have been treated with drugs, orthotics and referred to physical rehabilitation (physiotherapy and/or physical activity). Patients will be randomized into 2 groups of 76 and will go through pre-assessment with multidisciplinary team: Psychologist - assess cognitive ability; level of anxiety, and depression. Nutritionist - anthropometric parameters and diet quality. Social Worker - Level of education, religion, autonomy and mobility capacity to the hospital. Physiotherapist - range of motion, pain, function and quality of life. Occupational Therapy - range of motion and strength. Physical Educator - level of physical activity and functional capacity. Orthopaedic - additional examinations, disease classification, orthotics, report to Social Security and Traffic Department, evaluation questionnaires (SF 36, VAS, WOMAC, LEQUESNE), referral to physical therapy, physical activity and inform consent. A group will submitted to two interventions, with an interval of two months between each intervention. The control group will only make evaluations / consultations with all professional teams without classes for 2 years, then will attend the courses and will be followed by two more years. Interventions will be lectures and practices with the seven professional teams, covering the topic arthritis (orthopedic team), what is disease, being ill, and the role of the patient in the treatment (psychology) to obtain behavioral change. Lectures and practices with physical therapy and occupational therapy to show the importance of exercise in relieving symptoms (physical therapy), the importance of rest and proper ergonomics at home and at work (occupational therapy). The nutritionist shows proper alimentation. Lecture and practice with physical educator (showing the difference between the laber work and regular physical activity as well as the importance of strength exercises, resistance and stretching) and theoretical class with the social service by calling attention to the importance of leisure. After two months, the second intervention is made in order to verify the acquired concepts. Six months, 1, 2, 3 and 4 years after the first evaluation, the groups will be called to new multi evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with primary osteoarthritis of the knee,
* Classified as stages I to III of Kelgreen and Lawrence (KL), ie any degree of gonarthritis without obliteration of the joint space.
* With indication for clinical treatment of OA.

Exclusion Criteria:

* Patients with cognitive, psychiatric and neurological disorders or whose symptoms during the evaluation are related or significantly interfere in the functions of attention, memory, logical thinking, understanding and interaction with the group in order to hinder the assimilation of the given guidelines.

Missing classroom interventions

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Improvement in pain of patients with knee osteoarthritis by multi-professional care and education. (Visual Analogue Scale (VAS) and Womac) | 5 years
  Visual Analogue Scale (VAS) and Womac pain at 6 months, 1, 2, 3 and 4 years
Improvement in function of patients with knee osteoarthritis by multi-professional care and education. (testing and HAQ (Health Assessment Questionnaire )and DASH (Disabilities of the Arm, Shoulder And Hand questionnaires) | 5 years
  Lequesne, Womac, TUG (Timed Up and Go), FTSST ( Five Time Sit to Stand Test), Sit to Stand 30 Second Test, Palmar pressure force, Digital pinch strength, Range of motion (ROM) of the upper limbs (UL), Application of HAQ (Health Assessment Questionnaire )and DASH (Disabilities of the Arm, Shoulder And Hand questionnaires) at 6 months, 1, 2, 3 and 4 years
Improvement in percentage of body fat of patients with knee osteoarthritis by multi-professional care and education. (skinfolds measurements) | 5 years
  Nine skinfolds measurements at 6, 12, 24, 36 and 48 months
quality of life of patients with knee osteoarthritis by multi-professional care and education.. | 5 years
  SF-36 at 6, 12, 24, 36 and 48 months

SECONDARY OUTCOMES:
Evaluate increase physical activity of patients with knee osteoarthritis by multi-professional care and education. (Minutes per week of light, moderate or intense physical acitivity) | 5 years
  Minutes per week of light, moderate or intense physical acitivity
Evaluate changes in BMI of patients with knee osteoarthritis by multi-professional care and education. | 5 years
  By measuring height and weight at 6, 12, 24, 36 and 48 months.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia U Rezende, MD. PhD, Principal Investigator — Department of Orthopedics and Traumatology - Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo
Locations (2):
- Brazil (2):
  - Instituto de Ortopedia e Traumatologia do Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Instituto de Ortopedia e Traumatologia - HCFMUSP, São Paulo

REFERENCES:
- [Background] Lane NE, Brandt K, Hawker G, Peeva E, Schreyer E, Tsuji W, Hochberg MC. OARSI-FDA initiative: defining the disease state of osteoarthritis. Osteoarthritis Cartilage. 2011 May;19(5):478-82. doi: 10.1016/j.joca.2010.09.013. Epub 2011 Mar 23. PMID 21396464
- [Background] Woolf AD, Pfleger B. Burden of major musculoskeletal conditions. Bull World Health Organ. 2003;81(9):646-56. Epub 2003 Nov 14. PMID 14710506
- [Background] WHO Scientific Group on the Burden of Musculoskeletal Conditions at the Start of the New Millennium. The burden of musculoskeletal conditions at the start of the new millennium. World Health Organ Tech Rep Ser. 2003;919:i-x, 1-218, back cover. PMID 14679827
- [Background] Kwok WY, Vliet Vlieland TP, Rosendaal FR, Huizinga TW, Kloppenburg M. Limitations in daily activities are the major determinant of reduced health-related quality of life in patients with hand osteoarthritis. Ann Rheum Dis. 2011 Feb;70(2):334-6. doi: 10.1136/ard.2010.133603. Epub 2010 Nov 15. PMID 21081529
- [Background] Dawson J, Linsell L, Zondervan K, Rose P, Randall T, Carr A, Fitzpatrick R. Epidemiology of hip and knee pain and its impact on overall health status in older adults. Rheumatology (Oxford). 2004 Apr;43(4):497-504. doi: 10.1093/rheumatology/keh086. Epub 2004 Feb 3. PMID 14762225
- [Background] Dixon T, Shaw M, Ebrahim S, Dieppe P. Trends in hip and knee joint replacement: socioeconomic inequalities and projections of need. Ann Rheum Dis. 2004 Jul;63(7):825-30. doi: 10.1136/ard.2003.012724. PMID 15194578
- [Background] Mahomed NN, Barrett J, Katz JN, Baron JA, Wright J, Losina E. Epidemiology of total knee replacement in the United States Medicare population. J Bone Joint Surg Am. 2005 Jun;87(6):1222-8. doi: 10.2106/JBJS.D.02546. PMID 15930530
- [Background] Blagojevic M, Jinks C, Jeffery A, Jordan KP. Risk factors for onset of osteoarthritis of the knee in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2010 Jan;18(1):24-33. doi: 10.1016/j.joca.2009.08.010. Epub 2009 Sep 2. PMID 19751691
- [Background] Jorgensen KT, Pedersen BV, Nielsen NM, Hansen AV, Jacobsen S, Frisch M. Socio-demographic factors, reproductive history and risk of osteoarthritis in a cohort of 4.6 million Danish women and men. Osteoarthritis Cartilage. 2011 Oct;19(10):1176-82. doi: 10.1016/j.joca.2011.07.009. Epub 2011 Jul 27. PMID 21835256
- [Background] Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden NK, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis: part III: Changes in evidence following systematic cumulative update of research published through January 2009. Osteoarthritis Cartilage. 2010 Apr;18(4):476-99. doi: 10.1016/j.joca.2010.01.013. Epub 2010 Feb 11. PMID 20170770
- [Derived] Rodrigues da Silva JM, de Rezende MU, Spada TC, da Silva Francisco L, Sabine de Farias FE, Clemente da Silva CA, Cernigoy CHA, Greve JMD, Ciolac EG. Educational program promoting regular physical exercise improves functional capacity and daily living physical activity in subjects with knee osteoarthritis. BMC Musculoskelet Disord. 2017 Dec 27;18(1):546. doi: 10.1186/s12891-017-1912-7. PMID 29282054
- See also: POF 2008-2009: desnutrição cai e peso das crianças brasileiras ultrapassa padrão internacional — http://saladeimprensa.ibge.gov.br/noticias?busca=1&id=1&idnoticia=1699&t=pof-20082009-desnutricao-cai-peso-criancas-brasileiras-ultrapassa-padrao-internacional&view=noticia
- See also: PARQVE-Project Arthritis Recovering Quality of Life by Means of Education Short-term Outcome in a Randomized Clinical Trial — https://www.omicsonline.org/peer-reviewed/parqveproject-arthritis-recovering-quality-of-life-by-means-of-education-shortterm-outcome-in-a-randomized-clinical-trial-20432.html